CLINICAL TRIAL: NCT00518414
Title: The Evaluation of Cow Milk-Based Formulas - Study A
Brief Title: The Evaluation of Cow Milk-Based Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 3378
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Term Infants
Keywords: infant, formula, LC PUFA
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Marketed infant formula with DHA and ARA (Active Comparator): Marketed milk-based infant formula containing docosahexaenoic acid (DHA) and arachidonic acid (ARA)
  Interventions: Other: Marketed infant formula with DHA and ARA
- Milk-based infant formula with DHA and ARA (Experimental): Experimental milk-based infant formula containing docosahexaenoic acid (DHA) and arachidonic acid (ARA)
  Interventions: Other: Milk-based infant formula with DHA and ARA
- Milk-based formula with DHA, ARA, prebiotics (Experimental): Experimental milk-based infant formula containing docosahexaenoic acid (DHA) and arachidonic acid (ARA) and prebiotic blend
  Interventions: Other: Milk-based formula with DHA, ARA, prebiotics

INTERVENTIONS:
Other: Marketed infant formula with DHA and ARA
  Arms: Marketed infant formula with DHA and ARA
Other: Milk-based infant formula with DHA and ARA
  Arms: Milk-based infant formula with DHA and ARA
Other: Milk-based formula with DHA, ARA, prebiotics
  Arms: Milk-based formula with DHA, ARA, prebiotics

SUMMARY:
Infants will be fed infant formula and blood drawn to measure fatty acid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infant
* 10 to 18 days of age

Exclusion Criteria:

* Breast fed infants
* Infants with formula intolerance

Ages: 10 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell (RBC) ARA and DHA | 120 Days of age

SECONDARY OUTCOMES:
Phospholipid fatty acids, tolerance | 120 Days of age

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Berseth, M.D., Study Director — Mead Johnson Nutritionals
Locations (9):
- United States (9):
  - Birmingham Pediatric Group, Birmingham, Alabama
  - Southlake Pediatrics, Birmingham, Alabama
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Children's Medical Association, Tamarac, Florida
  - Welborn Clinic, Evansville, Indiana
  - The Center for Human Nutrition, Omaha, Nebraska
  - Holston Medical Group, Kingsport, Tennessee
  - DCOL Center for Clinical Research, Longview, Texas
  - Northwood Pediatrics, The Woodlands, Texas